CLINICAL TRIAL: NCT00020150
Title: Phase I Trial and Pharmacokinetic Study of Temozolomide and O6-Benzylguanine in Childhood Solid Tumors
Brief Title: Temozolomide and O6-benzylguanine in Treating Children With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067880; NCI-00-C-0105I; NCI-237; NCT00005019 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2004-08

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Kidney Cancer; Liver Cancer; Neuroblastoma; Ovarian Cancer; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: recurrent childhood rhabdomyosarcoma; childhood craniopharyngioma; recurrent childhood brain tumor; recurrent neuroblastoma; recurrent childhood liver cancer; recurrent Wilms tumor and other childhood kidney tumors; childhood central nervous system germ cell tumor; recurrent osteosarcoma; unspecified childhood solid tumor, protocol specific; childhood germ cell tumor; recurrent childhood soft tissue sarcoma; childhood oligodendroglioma; childhood choroid plexus tumor; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent childhood visual pathway and hypothalamic glioma; previously treated childhood rhabdomyosarcoma; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent childhood ependymoma; childhood teratoma; childhood malignant testicular germ cell tumor; childhood extragonadal germ cell tumor; childhood malignant ovarian germ cell tumor; recurrent childhood malignant germ cell tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Kidney Neoplasms; Liver Neoplasms; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Wilms Tumor; Osteosarcoma; Oligodendroglioma; Choroid Plexus Neoplasms; Astrocytoma; Medulloblastoma; Optic Nerve Glioma; Neuroectodermal Tumors, Primitive, Peripheral; Familial ependymoma; Teratoma; Testicular Neoplasms; Ovarian Germ Cell Cancer | interventions — O(6)-benzylguanine; Temozolomide

INTERVENTIONS:
Drug: O6-benzylguanine
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining temozolomide and O6-benzylguanine in treating children who have solid tumors that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of temozolomide administered with a biologically active dose of O6-benzylguanine (O6-BG) in children with refractory solid tumors.
* Determine the dose-limiting toxicity and the toxicity profile of this combination in these patients.
* Assess the plasma pharmacokinetics of O6-BG and its active metabolite, 8-oxo-O6-BG, in these patients.
* Assess the plasma pharmacokinetics of this combination in these patients.
* Correlate levels of alanine-glyoxylate aminotransferase in peripheral blood mononuclear cells with the degree of hematologic toxicity of this combination in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive O6-benzylguanine (O6-BG) IV over 1 hour followed 30 minutes later by oral temozolomide daily for 5 days. Treatment continues every 28 days for up to 12 courses in the absence of unacceptable toxicity or disease progression.

Sequential dose escalation of O6-BG is followed by sequential dose escalation of temozolomide. Cohorts of 3-6 patients receive escalating doses of O6-BG and temozolomide until the maximum tolerated dose (MTD) of each is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 6 patients experience dose-limiting toxicity.

Quality of life is assessed at baseline and prior to courses 1, 3, 6, 8, and 12.

PROJECTED ACCRUAL: A total of 21-48 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor refractory to standard therapy and for which no potentially curative therapy exists, including, but not limited to:

  * Rhabdomyosarcoma and other soft tissue sarcomas
  * Ewing's family of tumors
  * Osteosarcoma
  * Neuroblastoma
  * Wilms' tumor
  * Hepatic tumors
  * Germ cell tumors
  * Primary brain tumor
* Histological confirmation may be waived for brainstem or optic gliomas
* Measurable or evaluable disease
* Evidence of progressive disease on prior chemotherapy or radiotherapy or persistent disease after prior surgery

PATIENT CHARACTERISTICS:

Age:

* 21 and under

Performance status:

* ECOG 0-2

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Absolute granulocyte count greater than 1,500/mm^3
* Hemoglobin greater than 8 g/dL
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin normal
* SGPT less than 2 times upper limit of normal
* No significant hepatic dysfunction

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No significant cardiac dysfunction

Pulmonary:

* No significant pulmonary dysfunction

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow capsules
* No significant unrelated systemic illness that would preclude study (e.g., serious infections or organ dysfunction)
* No prior hypersensitivity to dacarbazine, temozolomide, or polyethylene glycol

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior colony-stimulating factors (e.g., filgrastim [G- CSF], sargramostim [GM-CSF], or epoetin alfa)
* At least 4 months since prior myeloablative therapy requiring bone marrow or stem cell transplantation
* No concurrent anticancer immunotherapy

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (4 weeks for nitrosoureas) and recovered
* Prior temozolomide allowed provided not administered within past 3 months, no severe toxicities experienced during prior course, and not given in combination with other agents designed to inactivate alanine-glyoxylate aminotransferase
* No other concurrent investigational or standard anticancer chemotherapy

Endocrine therapy:

* Concurrent corticosteroids for control of brain tumor-associated edema allowed provided on stable or decreasing dose for at least 1 week prior to study

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior limited-field radiotherapy
* At least 4 months since prior craniospinal irradiation, total body irradiation, or radiotherapy to more than half of the pelvis
* Recovered from prior radiotherapy
* No concurrent anticancer radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 4 weeks since other prior investigational therapy and recovered
* No other concurrent anticancer investigational agents

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Warren, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Meany HJ, Warren KE, Fox E, Cole DE, Aikin AA, Balis FM. Pharmacokinetics of temozolomide administered in combination with O6-benzylguanine in children and adolescents with refractory solid tumors. Cancer Chemother Pharmacol. 2009 Dec;65(1):137-42. doi: 10.1007/s00280-009-1015-8. Epub 2009 May 9. PMID 19430790
- [Result] Warren KE, Aikin AA, Libucha M, Widemann BC, Fox E, Packer RJ, Balis FM. Phase I study of O6-benzylguanine and temozolomide administered daily for 5 days to pediatric patients with solid tumors. J Clin Oncol. 2005 Oct 20;23(30):7646-53. doi: 10.1200/JCO.2005.02.0024. PMID 16234526